CLINICAL TRIAL: NCT00413920
Title: A Multicenter Randomized Open Label Study to Assess Efficacy and Safety of a Steroid Avoidance Regimen in Comparison to a Treatment With Steroids, in Combination With Enteric-coated Mycophenolate Sodium (EC-MPS) 2.16 g/d for 6 Weeks and Cyclosporine Microemulsion, in de Novo Adult Renal Transplant Recipients
Brief Title: Efficacy and Safety of Enteric-coated Mycophenolate Sodium and Cyclosporine in Combination With and Without Steroids, in Adult Renal Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080AFR05
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Results first posted 2011-02-07 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Renal Transplantation
Keywords: Steroids avoidance,; enteric-coated mycophenolate sodium (EC-MPS),; de novo renal transplantation
MeSH Terms: interventions — Mycophenolic Acid; Prednisone

ARMS (2):
- Without Steroids (Experimental): Patients received Enteric-coated Mycophenolate Sodium (EC-MPS), administered orally 2 times a day for 6 months. Patients also received cyclosporine and a dose of methylprednisolone immediately after transplantation, but did not subsequently receive oral corticosteroids for the remainder of the study.
  Interventions: Drug: Enteric-coated mycophenolate sodium (EC-MPS)
- With Steroids (Active Comparator): Patients received Enteric-coated Mycophenolate Sodium (EC-MPS), administered orally 2 times a day for 6 months. Patients also received cyclosporine and a dose of methylprednisolone immediately after transplantation, and subsequently continued to receive daily oral prednisone.
  Interventions: Drug: Enteric-coated mycophenolate sodium (EC-MPS); Drug: Prednisone

INTERVENTIONS:
Drug: Enteric-coated mycophenolate sodium (EC-MPS) — An initial dose of 1080 mg EC-MPS was administered immediately before transplantation. Then, during the first 6 weeks post-transplantation, EC-MPS was administered at a dose of 1080 mg twice a day 12 hours apart. From week 7 until the end of the study (month 6), EC-MPS was administered at standard dose of 720 mg twice a day.
  Other Names: Myfortic
Drug: Prednisone — Oral tablets
  Arms: With Steroids

SUMMARY:
This study will investigate the efficacy and safety of a steroid avoidance regimen in comparison with steroid treatment in combination with an initially higher dose of enteric-coated mycophenolate sodium (EC-MPS) and cyclosporine microemulsion in de novo renal transplant recipients. Patients will be randomly allocated to receive either EC-MPS or steroids in combination with EC-MPS. Patients of both treatment groups will receive monoclonal antibody induction therapy and a perioperative bolus of steroids and cyclosporine.

ELIGIBILITY:
Inclusion Criteria:

* Primary donor kidney transplant
* Panel reactive antibody (PRA) ≤ 20%

Exclusion Criteria:

* Multi-organ transplantation including dual kidneys or previous transplant with any other organ different from kidney
* Non-heart beating donor or kidney from a non-compatible donor

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- C.H.U. La Milétrie, Poitiers, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Without Steroids | With Steroids
Started | 112 | 110
Completed | 84 | 82
Not Completed | 28 | 28
Not completed — Adverse Event | 9 | 11
Not completed — Lack of Efficacy | 11 | 9
Not completed — Death | 3 | 5
Not completed — Graft Loss | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Without Steroids | With Steroids | Total
Number analyzed (Participants) | 112 | 110 | 222
Age Continuous [Mean (Standard Deviation); unit: years] | 51.0 (10.24) | 50.9 (11.91) | 51.0 (11.07)
Age, Customized [Number; unit: Participants]
  < 45 years | 33 | 25 | 58
  45-60 years | 56 | 58 | 114
  >= 60 years | 23 | 27 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 40 | 76
  Male | 76 | 70 | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Occurrence of Treatment Failures at 6 Months Post-transplantation
Description: Treatment failures defined as Biopsy Proven Acute Rejection (BPAR), graft loss, death or loss to follow-up. Only BPAR from other biopsies than the protocol defined biopsy at Month 3 are described. Acute rejection: an episode of acute renal dysfunction diagnosed as rejection on the basis of biopsy or clinical observations, treated with anti-rejection medication. BPAR: renal transplant biopsy finding of acute cellular or antibody mediated rejection. Graft loss: allograft will be presumed to be lost on the day the patient starts dialysis and is not able to subsequently be removed from dialysis.
Time Frame: 6 months post transplantation
Population: Intent-to-treat population
Measure: Number; unit: Number of participants
Arm/Group | Without Steroids | With Steroids
Number analyzed (Participants) | 112 | 110
Number of participants | 20 | 16

2. Secondary Outcome: The Number of Participants With BPAR, Clinical Acute Rejection (AR) and Treated AR at 6 Months
Description: If a participant experienced several BPAR, only the rejection with highest grade is taken into account. Only events that occurred before study treatment discontinuation are taken into account. Only BPAR from other biopsies than the protocol defined biopsy at Month 3 are described. Acute rejection: an episode of acute renal dysfunction diagnosed as rejection on the basis of biopsy or clinical observations, treated with anti-rejection medication. BPAR: renal transplant biopsy finding of acute cellular or antibody mediated rejection.
Time Frame: Month 6
Population: Intent-to-treat population
Measure: Number; unit: Number of participants
Arm/Group | Without Steroids | With Steroids
Number analyzed (Participants) | 112 | 110
Number of participants
  Biopsy Proven Acute Rejection | 13 | 8
  Graft Loss | 5 | 3
  Death | 2 | 5
  Loss to Follow-up | 0 | 0
  Acute Rejection | 37 | 21
  Treated Acute Rejection | 36 | 19

3. Secondary Outcome: Number of Participants With Treatment Failure, BPAR, Clinical Acute Rejection (AR) and Treated AR at 3 Months
Description: A treatment failure is a Biopsy Proven Acute Rejection (BPAR), a graft loss, a death, or a loss to follow-up. Only BPAR from other biopsies than the protocol defined biopsy at Month 3 are described. Acute rejection: an episode of acute renal dysfunction diagnosed as rejection on the basis of biopsy or clinical observations, treated with anti-rejection medication. BPAR: renal transplant biopsy finding of acute cellular or antibody mediated rejection. Graft loss: The allograft will be presumed lost on the day the patient starts dialysis and is not able to subsequently be removed from dialysis.
Time Frame: Month 3
Population: Intent-to-treat population
Measure: Number; unit: Number of participants
Arm/Group | Without Steroids | With Steroids
Number analyzed (Participants) | 112 | 110
Number of participants
  Treatment Failure | 17 | 8
  Biopsy Proven Acute Rejection | 10 | 5
  Graft Loss | 5 | 1
  Death | 2 | 2
  Loss to Follow-up | 0 | 0
  Acute Rejection | 32 | 19
  Treated Acute Rejection | 31 | 16

4. Secondary Outcome: Number of Participants With Subclinical Histological Rejections
Description: The number of participants with subclinical histological rejections was determined by renal biopsy screening at 3 months in 125 patients, providing adequate samples for 112 biopsies.
Time Frame: Month 3
Population: Intent-to-treat population on whom biopsies were performed at 3 months.
Measure: Number; unit: Number of participants
Arm/Group | Without Steroids | With Steroids
Number analyzed (Participants) | 59 | 66
Number of participants
  Sample quality inadequate | 7 | 6
  Subclinical rejection | 12 | 17
  Borderline lesions | 2 | 5
  BPAR | 10 | 12

5. Secondary Outcome: Number of Participants With Treatment Failure at 3 Months by Graft Recovery Status
Description: The number of participants with treatment failure defined as a Biopsy Proven Acute Rejection (BPAR), a graft loss, a death, or a loss to follow-up at 3 months by graft recovery status.
  Delayed graft function is defined as the need for dialysis within the first 7 days post-transplantation, excluding the first post-transplantation day.
  Slow graft function is defined as a serum creatinine value > 250 µmol/L at day 5.
Time Frame: Month 3
Population: Intent-to-treat population. N in the categories is the number of participants from the total population that fit into that category for each arm/group. For example: in the Delayed Graft Function category there were 25 participants in the Without steroid group and 24 participants in the With Steroid Group.
Measure: Number; unit: Number of participants
Arm/Group | Without Steroids | With Steroids
Number analyzed (Participants) | 112 | 110
Number of participants
  Delayed Graft Function [N= 25,24] | 8 | 4
  Slow Graft Function [N= 36,23] | 6 | 1
  Immediate Graft Function [N= 51,63] | 3 | 3

6. Secondary Outcome: Number of Participants Requiring Steroids in Non-steroid Treatment Group
Time Frame: Months 3 and 6
Measure: Number; unit: Number of participants
Arm/Group | Without Steroids
Number analyzed (Participants) | 112
Number of participants
  3 Months | 25
  6 Months | 20

ADVERSE EVENTS:
Arm/Group | Without Steroids | With Steroids
Serious Adverse Events (participants affected / at risk) | 72/112 | 69/110
Other Adverse Events (participants affected / at risk) | 104/112 | 107/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Without Steroids (N=112) | With Steroids (N=110)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemoglobinaemia (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 4
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 2
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 6
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Malabsorption (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 2 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 4
Asthenia (General disorders) | 3 | 0
Catheter site pain (General disorders) | 1 | 0
Chills (General disorders) | 5 | 3
Death (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Hyperthermia (General disorders) | 3 | 4
Inflammation (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 2 | 1
Pain (General disorders) | 0 | 1
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 10 | 10
Sudden death (General disorders) | 0 | 3
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 1
Kidney transplant rejection (Immune system disorders) | 1 | 1
Transplant rejection (Immune system disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 6 | 10
Diarrhoea infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Graft infection (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 2 | 1
Infected lymphocele (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 0
Mycotic aneurysm (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Perinephric abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 5 | 9
Pyelonephritis acute (Infections and infestations) | 3 | 1
Renal cyst infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 3
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 4
Viral infection (Infections and infestations) | 1 | 1
Wound abscess (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 3 | 4
Drug toxicity (Injury, poisoning and procedural complications) | 2 | 2
Graft complication (Injury, poisoning and procedural complications) | 1 | 2
Graft dysfunction (Injury, poisoning and procedural complications) | 8 | 8
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 3 | 0
Perinephric collection (Injury, poisoning and procedural complications) | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 2
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Renal injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 5 | 0
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Venous injury (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 10 | 8
Creatinine urine increased (Investigations) | 1 | 0
Immunosuppressant drug level increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1
Overweight (Metabolism and nutrition disorders) | 0 | 1
Sodium retention (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Drug abuse (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Bladder necrosis (Renal and urinary disorders) | 0 | 1
Detrusor sphincter dyssynergia (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Nephritis (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Pyelocaliectasis (Renal and urinary disorders) | 1 | 1
Renal aneurysm (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal artery thrombosis (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 2 | 2
Renal failure acute (Renal and urinary disorders) | 12 | 10
Renal impairment (Renal and urinary disorders) | 3 | 3
Renal infarct (Renal and urinary disorders) | 0 | 1
Renal ischaemia (Renal and urinary disorders) | 0 | 1
Renal tubular disorder (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0
Ureteral necrosis (Renal and urinary disorders) | 1 | 0
Ureteric dilatation (Renal and urinary disorders) | 2 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 5 | 2
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0
Urinoma (Renal and urinary disorders) | 1 | 2
Urogenital disorder (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Catheter removal (Surgical and medical procedures) | 0 | 1
Nephrectomy (Surgical and medical procedures) | 1 | 0
Nephrostomy tube removal (Surgical and medical procedures) | 0 | 1
Transurethral prostatectomy (Surgical and medical procedures) | 0 | 1
Venous ligation (Surgical and medical procedures) | 1 | 0
Angiosclerosis (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0
Axillary vein thrombosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Extrinsic vascular compression (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 3 | 2
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 3 | 5
Orthostatic hypotension (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Without Steroids (N=112) | With Steroids (N=110)
Anaemia (Blood and lymphatic system disorders) | 60 | 56
Leukopenia (Blood and lymphatic system disorders) | 21 | 12
Abdominal pain (Gastrointestinal disorders) | 12 | 6
Aphthous stomatitis (Gastrointestinal disorders) | 4 | 6
Constipation (Gastrointestinal disorders) | 17 | 17
Diarrhoea (Gastrointestinal disorders) | 15 | 16
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 7
Gingival hypertrophy (Gastrointestinal disorders) | 8 | 8
Oedema peripheral (General disorders) | 27 | 27
Pain (General disorders) | 15 | 13
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 8
Bronchitis (Infections and infestations) | 5 | 8
Cytomegalovirus infection (Infections and infestations) | 9 | 16
Urinary tract infection (Infections and infestations) | 34 | 39
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 8 | 9
Graft dysfunction (Injury, poisoning and procedural complications) | 16 | 18
Blood phosphorus decreased (Investigations) | 4 | 6
Acidosis (Metabolism and nutrition disorders) | 8 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 10 | 11
Dyslipidaemia (Metabolism and nutrition disorders) | 10 | 21
Fluid retention (Metabolism and nutrition disorders) | 9 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 30 | 31
Hyperkalaemia (Metabolism and nutrition disorders) | 19 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 17
Tremor (Nervous system disorders) | 10 | 7
Insomnia (Psychiatric disorders) | 20 | 18
Haematuria (Renal and urinary disorders) | 8 | 7
Proteinuria (Renal and urinary disorders) | 6 | 9
Hypertension (Vascular disorders) | 20 | 17
Lymphocele (Vascular disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.